CLINICAL TRIAL: NCT07200245
Title: Cardiovascular Complications After Adrenalectomy for Pheochromocytoma and Non-secreting Tumors - A Prospective Observational Multicenter European Study (HEMODYNAMICS)
Brief Title: Cardiovascular Complications After Adrenalectomy for Pheochromocytoma and Non-secreting Tumors
Acronym: HEMODYNAMICS
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Eurocrine Council (Unknown); European Society of Endocrine Surgery (ESES) (Unknown)
Responsible Party: Principal Investigator, Laurent BRUNAUD, Clinical professor (PUPH), Central Hospital, Nancy, France
Other Study IDs: 8372 - Endocrine Tumour Base
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pheochromocytoma; Cardiovascular Complication; Adrenal Incidentaloma
MeSH Terms: conditions — Pheochromocytoma; Adrenal incidentaloma | interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pheochromocytoma: adrenalectomy for pheochromocytoma
  Interventions: Other: adrenalectomy
- non-secreting tumor: adrenalectomy for non-secreting tumor (incidentaloma)
  Interventions: Other: adrenalectomy

INTERVENTIONS:
Other: adrenalectomy — adrenalectomy for pheochromocytoma and non-secreting tumor (incidentaloma)

SUMMARY:
Pheochromocytoma is an adrenomedullary chromaffin cell tumour that releases catecholamines. Adverse cardiovascular events are considered the main cause of morbidity and mortality in patients with pheochromocytoma. Consequently, preoperative medical preparations using alpha-blockers or other antihypertensive drugs and the control of hemodynamic instability during adrenalectomy for pheochromocytoma are recommended by guidelines to prevent vasoconstriction, perioperative cardiovascular complications, and the risk of death. However, the definition of a catecholamine-induced hypertensive crisis in patients with pheochromocytoma has only recently been validated by an international consortium as the occurrence of systolic/diastolic blood pressure >180/120 mmHg1. Limitations of published studies include small sample sizes, and single institution analysis. Some studies have reported substantial variability in the management of pheochromocytomas, with the use of routine preoperative medical preparation varying from 49% to 100%, whereas others have questioned the utility of this preparation for postoperative cardiovascular complications. The aim of this study was to evaluate pan-European practices in terms of specific preoperative medical preparation before surgery and to identify risk factors for postoperative cardiovascular complications 30 days after adrenalectomy for pheochromocytoma and non-secreting tumors (indication for surgery = " excluding malignancy ").

The EUROCRINE® registry offers a valuable opportunity to assess clinical practices for preoperative medical preparation and the morbidity linked to adrenalectomy for pheochromocytoma and non-secreting tumors. This prospective study aims to refine surgical protocols and inform updates to existing guidelines, thereby advancing the management of adrenalectomy for pheochromocytoma.

DETAILED DESCRIPTION:
The investigators propose a prospective, observational, multicenter, multinational study based on the EUROCRINE® registry. The study will use the my-EUROCRINE® module to add study-specific variables for patients included in the study protocol. Medical centers that transfer data to the EUROCRINE® registry will be invited to participate in this project. Patients with pheochromocytoma and non-secreting tumor (corresponding to patients with indication for surgery = " excluding malignancy ") will be included.

All patients included will undergo a preoperative biological assessment (blood, urine, or not performed), an assessment of the dosage and duration of preoperative medical preparation using alpha-blockers (or not performed), an assessment of all intraoperative hypertensive and hypotensive crises (duration of all episodes defined according to validated criteria), and an assessment of cardiovascular complications at day 30 using a predefined definition of nine cardiovascular events.

Consecutive patient enrolment is necessary to accurately reflect real clinical conditions. The standard variables are recorded as usual, with the addition of extra-variables (using My Eurocrine module) and detailed in the case report form (CRF).

For defining intraoperative hypertensive episode(s), the investigators opted to utilize the established Nazari et al. definition published in 2023 (> 180 mmHg for systolic blood pressure and/or > 120 mmHg for diastolic blood pressure)1. For defining intraoperative hypotensive episode(s), the investigators used the Sessler and al. published definition in 2019 (mean arterial pressure < 65 mmHg)(POQI consensus)3. For these two intraoperative criteria, the total duration (in minutes from induction to discharge from the operating room) of the episodes will be collected at the end of the adrenalectomy in collaboration with the anesthesia team.

For defining intraoperative cardiovascular complications and at 30 days after adrenalectomy, the investigators used the definition by Beattie et al.2, which corresponds to the presence of one or more of the nine clearly defined following events: myocardial infarction (MI), myocardial injury, cardiovascular death, non-fatal cardiac arrest (NFCA), coronary revascularization (CR), major adverse cardiac events (cardiac death or MI or CR or NFCA), pulmonary embolism, deep vein thrombosis, and atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adrenalectomy for pheochromocytoma
* Patients undergoing adrenalectomy for non-secreting tumors. Patients with non-secreting tumors are those with indication for adrenalectomy in the Eurocrine database corresponding to " excluding malignancy ".

Exclusion Criteria:

* Children and minors (<18 years).
* Pregnant women.
* Patients with other indication for adrenalectomy in Eurocrine (i.e. Adrenocortical cancer, Cushing, Primary aldosteronism, Metastasis).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, observational, multicenter, multinational study based on the EUROCRINE® registry. The study will use the my-EUROCRINE® module to add study-specific variables for patients included in the study protocol. Centers that transfer data to the EUROCRINE® registry will be invited to participate in this project. Patients with pheochromocytoma and non-secreting tumor (corresponding to patients with indication for surgery = " excluding malignancy ") will be included.
Sampling Method: Probability Sample
Enrollment: 522 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiovascular complications at postoperative day 30 | 30 days
  cardiovascular complications at postoperative day 30 among the following cardiovascular events: myocardial infarction (MI), myocardial injury, cardiovascular death, non-fatal cardiac arrest (NFCA), coronary revascularization (CR), major adverse cardiac events (cardiac death or MI or CR or NFCA), pulmonary embolism, deep vein thrombosis, and atrial fibrillation.

SECONDARY OUTCOMES:
Intraoperative hypertensive episodes | from induction of general anesthesia until discharge from the operating room
  duration of all intraoperative blood pressure episode(s) > 180 mmHg systolic and/or > 120 mmHg diastolic between induction and discharge from the operating room (duration in minutes)
Intraoperative hypotensive episodes | from induction of general anesthesia until discharge from the operating room
  duration of all intraoperative mean arterial pressure episode(s) below 65 mmHg between induction and discharge from the operating room (duration in minutes).

CONTACTS AND LOCATIONS:
Overall Officials: laurent BRUNAUD, MD, PhD, Principal Investigator — University of Lorraine, CHRU Nancy,

IPD SHARING:
Plan to Share IPD: No